CLINICAL TRIAL: NCT04123678
Title: Impact of an Artificial Intelligence Platform (DERM) on the Healthcare Resource Utilisation (HRU) Needed to Diagnose Skin Cancer When Used as Part of a United Kingdom-based Teledermatology Service
Brief Title: DERM Health Economics Study
Status: Completed | Type: Observational
Sponsor: Skin Analytics Limited (Industry)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: DERM-005
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Melanoma; Non-melanoma Skin Cancer
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All: Patients attending a Medical Photography facility with at least 1 suspicious skin lesion will be approached to participate in the study. Participants will have an additional macro and dermoscopic image of each suspicious skin lesions suitable for photography. Photographs will be taken by a healthcare professional using an iPhone XR smart phone camera with a DL1 dermoscopic lens attachment. The images will be encrypted and electronically transmitted to Skin Analytics' cloud servers for analysis by DERM. The suspected diagnosis determined by DERM will be compared with dermatologist review and histologically confirmed diagnosis, where obtained. Healthcare resource utilization information and patient satisfaction data will also be collected
  Interventions: Device: Deep Ensemble for the Recognition of Malignancy (DERM)

INTERVENTIONS:
Device: Deep Ensemble for the Recognition of Malignancy (DERM) — AI-based decision support tool

SUMMARY:
This study aims to provide an initial assessment of the potential impact DERM could have on the number of onward referrals for a face to face dermatologist review and/or biopsy from a teledermatology-based service, and to improve the understanding of the patient pathways that exist.

DETAILED DESCRIPTION:
DERM, an Artificial Intelligence (AI)-based diagnosis support tool, has been shown to be able to accurately identify melanoma, non-melanoma skin cancers (NMSC) and other conditions from historical images of suspicious skin lesions (moles).

This study aims to establish whether the use of DERM in the patient pathway could reduce the number of unnecessary referrals to dermatologist review and/or biopsy.

Suspicious skin lesions that are due to be photographed for a dermatologist to review, will have two additional photographs taken using a commonly available smart phone camera with and without a specific lens attachment. The images will be analysed by DERM, and the results compared to the clinician's diagnosis (all lesions) and histologically-confirmed diagnosis (any lesion that is biopsied).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study,
* Male or Female, aged 18 years or above,
* Has at least one suspicious skin lesion which is being photographed as part of Standard of Care (SoC),
* In the Investigators opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients attending Medical Photography for imaging of at least 1 suspicious skin lesion. Patients may have been referred to the teledermatology service or for imaging for monitoring purposes from the dermatology clinic or for virtual teledermatology review.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Referral rate | Study completion, on average 5 days
  The rate of unnecessary referrals for a face to face dermatologist review for the same detection rate between standard of care and DERM of lesions reviewed by teledermatology or DERM

SECONDARY OUTCOMES:
Sensitivity of DERM on biopsied lesions | Study completion, on average 5 days
  Sensitivity of DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Specificity of DERM on biopsied lesions | Study completion, on average 5 days
  Specificity of DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
False positive rate of DERM on biopsied lesions | Study completion, on average 5 days
  False positive rate of DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
False negative rate of DERM on biopsied lesions | Study completion, on average 5 days
  False negative rate of DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Positive predictive value of DERM on biopsied lesions | Study completion, on average 5 days
  Positive predictive value of DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Number needed to biopsy by DERM on biopsied lesions | Study completion, on average 5 days
  Number needed to biopsy by DERM on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Sensitivity of teledermatologists on biopsied lesions | Study completion, on average 5 days
  Sensitivity of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Specificity of teledermatologists on biopsied lesions | Study completion, on average 5 days
  Specificity of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
False positive rate of teledermatologists on biopsied lesions | Study completion, on average 5 days
  False positive rate of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
False negative rate of teledermatologists on biopsied lesions | Study completion, on average 5 days
  False negative rate of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Positive predictive value of teledermatologists on biopsied lesions | Study completion, on average 5 days
  Positive predictive value of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Negative predictive value of teledermatologists on biopsied lesions | Study completion, on average 5 days
  Negative predictive value of teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Number needed to biopsy by teledermatologists on biopsied lesions | Study completion, on average 5 days
  Number needed to biopsy by teledermatologists on biopsied lesions, using histopathological confirmed diagnosis as gold-standard
Sensitivity of DERM to identify benign conditions | Study completion, on average 5 days
  Sensitivity of DERM to identify benign conditions, using clinical diagnosis as gold-standard
Specificity of DERM to identify benign conditions | Study completion, on average 5 days
  Specificity of DERM to identify benign conditions, using clinical diagnosis as gold-standard
False positive rate of DERM to identify benign conditions | Study completion, on average 5 days
  False positive of DERM to identify benign conditions, using clinical diagnosis as gold-standard
False negative rate of DERM to identify benign conditions | Study completion, on average 5 days
  False negative rate of DERM to identify benign conditions, using clinical diagnosis as gold-standard
Positive predictive value of DERM to identify benign conditions | Study completion, on average 5 days
  Positive predictive of DERM to identify benign conditions, using clinical diagnosis as gold-standard
Negative predictive value of DERM to identify benign conditions | Study completion, on average 5 days
  Negative predictive value of DERM to identify benign conditions, using clinical diagnosis as gold-standard
Number needed to refer by DERM to identify benign conditions | Study completion, on average 5 days
  Number needed to refer by DERM to identify benign conditions, using clinical diagnosis as gold-standard
Concordance of DERM result with clinical diagnosis | Study completion, on average 5 days
  Concordance of DERM result with clinical diagnosis
Percent of patients attending teledermatology by referral route | Study completion, on average 5 days
  Percentage of patients referred to teledermatology through 2-week wait referral, general referral, direct to teledermatology, routine follow-up (etc) referral routes
Time taken from general practitioner (GP) referral to diagnosis | Study completion, on average 5 days
  Time taken (days) from GP referral to either histopathology-confirmed or clinical diagnosis
Estimated cost impact associated with introducing DERM into the patient pathway | Study completion, on average 5 days
  The cost of the number of referrals for face to face dermatologist review and/or biopsy that would have been saved / charged if DERM had been used to decide whether to refer the patient onwards
Proportion of images submitted to DERM that cannot be analysed | Study completion, on average 5 days
  Proportion of images submitted to DERM that cannot be analysed
Patient satisfaction survey | Study completion, on average 5 days
  Patient feedback on their experience of the service. Patients will rate whether they agree, or don't agree, with statements that assess their acceptance of having a computer involved in their diagnosis pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Research to improve or test the performance of DERM only allowed in consent

REFERENCES:
- [Derived] Marsden H, Kemos P, Venzi M, Noy M, Maheswaran S, Francis N, Hyde C, Mullarkey D, Kalsi D, Thomas L. Accuracy of an artificial intelligence as a medical device as part of a UK-based skin cancer teledermatology service. Front Med (Lausanne). 2024 Mar 22;11:1302363. doi: 10.3389/fmed.2024.1302363. eCollection 2024. PMID 38585154